CLINICAL TRIAL: NCT01305980
Title: Phase Ⅱ,Open Label Clinical Trial to Investigate Safety and Efficacy of SB Injection in Patients With Advanced and Metastatic Colorectal Cancer
Brief Title: Evaluating the Safety and Efficacy of SB Injection in Patients With Advanced or Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SBPharmaceutical IND, Co., LTD (Industry)
Responsible Party: Lee Dong-heum / executive director, SBPharmaceutical IND, Co., LTD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB injection-C002
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB injection — Infusion SBinjection of 21.87ml/m^2, IV route, 24times for 4 months

SUMMARY:
The purpose of this study is to determine efficacy of SB injection in Colorectal Cancer.

DETAILED DESCRIPTION:
All eligible patients will receive SB injection therapy for 6 cycles (14~21 days for each cycle). Efficacy will be evaluated every 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18years or over
* Patients who had failed more than 1 cycle of standard therapy with advanced or metastatic stage and with measurable lesions
* Life expectancy >/= 5 months
* Not available to any of resectable surgery or radiotherapy
* Patients with adequate organ(e.g. heart, kidney, liver)and bone marrow function, as defined by

  1. Absolute neutrophil count >/= 1.0 x 10^9/L, Platelet count >/= 75 x 10^9/L
  2. Total bilirubin < 2.0 mg/dL
  3. Aspartate Aminotransferase and/or Aspartate Aminotransferase < 5 x Upper Limit Normal
  4. creatinine < 2 x Upper Limit Normal
* ECOG status 0 to 2
* Female volunteers admitted to the study must be using a reliable means of contraception and must have a negative blood or urine pregnancy test at least 7days ago
* Patients or their legal representatives who have signed the informed consent form.

Exclusion Criteria:

* Have inflammatory bowel diseases
* Have severe diarrhea or ileus
* Previous total colectomy
* Have ileostomy
* Known brain or spinal cord metastases
* Patients who have received chemotherapy within the previous 4 weeks
* Patients who have received radiotherapy related tp colorectal cancer within 4weeks
* Patients who have participated in other clinical study within the previous 4weeks
* Pregnancy or lactation period
* Human Immunodeficiency Virus antibody (+)
* Have active infection or serious concomitant systemic disorder incompatible with the study
* Clinically hypertension or diabetes mellitus not well controlled with medication
* Clinically significant cardiac disease(congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction
* Presence or history of malignancy other than colorectal cancer within 5years
* Have severe Neurologic or psychological disorder
* Patients who have history of allergy with this investigational drug(SB injection)
* Obvious cognitive or physical impairment that would prevent participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Evaluating Tumor Response Rate | 4 months

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 4 months
evaluate patient's performance by measuring Eastern Cooperative Oncology Group scale | 4 months
Determine duration of response rate by measuring time to progression | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong-oon Shin, Prof, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, Jung-gu, South Korea

REFERENCES:
- See also: SBP — http://www.sbp.com/